CLINICAL TRIAL: NCT04792684
Title: Collection of Samples From the United States Population for Optimization and Evaluation of Colorectal Cancer (CRC) Plasma Circulating Free-DNA (cfDNA) Marker Panel Performance ("USOPTIVAL")
Brief Title: Collection of Samples USOPTIVAL Study
Status: Recruiting | Type: Observational
Sponsor: Universal Diagnostics (Industry)
Responsible Party: Sponsor
Other Study IDs: CRC-US-001
Record Dates: First submitted 2021-03-08; First posted 2021-03-11 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Colorectal Cancer (CRC); Advanced Adenomas (AA)
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 40 ml of blood at the study visit processed for plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Arm A.: Subjects that have a suspected advanced adenoma or have been newly diagnosed with CRC still not resected and scheduled for surgery
  Interventions: Diagnostic Test: Optimization of Plasma Circulating Free-DNA (cfDNA) Marker Panel
- Arm B: Subjects at average-risk for CRC and scheduled for CRC screening colonoscopy
  Interventions: Diagnostic Test: Optimization of Plasma Circulating Free-DNA (cfDNA) Marker Panel

INTERVENTIONS:
Diagnostic Test: Optimization of Plasma Circulating Free-DNA (cfDNA) Marker Panel — Evaluate the performance of a preliminary panel of biomarkers

SUMMARY:
A prospective multi-center observational study. The study will enroll eligible subjects from the United States to optimize the biomarker panel and evaluate the performance of a cfDNA marker panel selected by the Sponsor for CRC and advanced adenoma detection.

DETAILED DESCRIPTION:
This study is designed to prospectively collect blood samples and clinical data from subjects that have a suspected advanced adenoma or have been newly diagnosed with CRC scheduled for resection surgery, as well as subjects who are at average-risk of colorectal cancer and who are scheduled for routine colonoscopy examination.

Subjects interested in participation and who meet inclusion criteria and provide written informed consent will be enrolled in the study. By accepting participation in the study, subjects will consent to provide up to 40 ml of blood at the study visit.

ELIGIBILITY:
Inclusion Criteria:

Arm A:

1. Must be 45-84 years of age.
2. Must have a suspected advanced adenoma or be newly diagnosed with CRC, still not resected, and scheduled for surgery.
3. Able to comprehend, sign, and date the written informed consent document.

Arm B:

1. Must be 45-84 years of age.
2. Able and willing to undergo a standard-of-care screening colonoscopy within 60 days.
3. Able to comprehend, sign, and date the written informed consent document.

Exclusion Criteria:

Arm A Only:

1. Subject with curative biopsy during colonoscopy.

Arm B Only:

1. Subjects with positive FIT Test results in the 6 months preceding enrollment.
2. Subject has a current diagnosis of cancer.

Arms A & B:

1. Subject has a personal history of aerodigestive or digestive tract cancers.
2. Subjects having undergone previous partial surgical removal of one or more portions of their colon due to a reason other than colorectal cancer.
3. Has a known diagnosis or personal history of any of the following high-risk indications for colorectal cancer:

   1. Inflammatory bowel disease (IBD) including chronic ulcerative colitis (CUC) and Crohn's disease.
   2. Familial adenomatous polyposis ("FAP", including attenuated FAP).
   3. Hereditary non-polyposis colorectal cancer syndrome ("HNPCC" or "Lynch Syndrome").
   4. Serrated polyposis syndrome
   5. 2 first-degree relatives (e.g., parents, siblings, and offspring) who have been diagnosed with colon cancer.
   6. One first-degree relative with CRC diagnosed before the age of 60.
4. A significant disease which, in the Investigator's opinion, would exclude the subject from the study.
5. Legal incapacity or limited mental capacity.
6. Medical or psychological conditions that would not permit the subject to complete the study or sign informed consent.
7. The patient has a known or documented previous or current medical history of infectious diseases that can be transmitted through blood (E.g. Hepatitis, HIV, etc.), including patients that have been treated, are currently being treated, or have not been treated for that conditions.
8. The patient is known to be pregnant when recruited or during her participation in the study.

Ages: 45 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Two cohorts of patients aged between 45 and 84, who have a suspected advanced adenoma or have been newly diagnosed with CRC, still not resected and scheduled for surgery, and patients who are at average risk of developing colorectal cancer, scheduled for a standard-of-care screening colonoscopy.
  Subjects will be considered enrolled after understanding and signing the ICF and a determination is made by the Investigator that the subject is eligible to participate according to the inclusion/exclusion criteria.
  Enrollment will be stopped when a sufficient number of confirmed cases of colorectal cancer, advanced adenomas, and matching control subjects have been enrolled. Under the current assumptions, 1,200 subjects will need to be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 1300 (Estimated)
Dates: Start 2020-12-30 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Samples Collected for Plasma Circulating Free-DNA (cfDNA) Marker Testing | Within 12 months of sample collection
  Samples Collected for Testing

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Precision Recearch Institute, Chula Vista, California
  - Precision Research Institute, San Diego, California
  - Medical Associates Research Group, San Diego, California
  - Clinical Research of California, Walnut Creek, California
  - Center for Gastrointestinal Disorders, Hollywood, Florida
  - Lakeland Regional Cancer Center, Lakeland, Florida
  - Springfield Clinic, Springfield, Illinois
  - Ochsner Clinic, New Orleans, Louisiana
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mid Hudson Medical Research, New Windsor, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Frontier Clinical Research, Uniontown, Pennsylvania
  - Clinical Trials Network, Union City, Tennessee
  - Vilo Research Group, Houston, Texas
  - Gastroenterology Consultants of SW Virginia, Raonoke, Virginia

IPD SHARING:
Plan to Share IPD: No